CLINICAL TRIAL: NCT05832866
Title: Effect of Clinic-based and Tele-monitored Home-based Intervention on Pain Intensity, Function and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Clinic-based and Tele-monitored Home-based Intervention in Patients With Knee OA
Acronym: CB&HMInKOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Professor, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ojoawo23/01
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Pain intensity; Functioning; Health Related Quality of Life; Tele-monitoring
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: There were two groups, one with clinical based and the other with telemonitored home based. The two groups received thera band exercises of isometric contractions. The clinical based at the hospital, and the home based at home but being monitored by researcher with phone call.
Who Masked: Participant
Masking Description: There was no masking in the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Based Isometric contraction strengthening Exercises using Thera band" CBG (Experimental): Participants underwent strengthening exercises to the quadriceps and harmstring using thera band at the hospital. The band was attached around the ankle for strengthening of the quadriceps and hamstring muscles using isometric muscle contraction using a standard protocol. The patient performed four sets of eight repetitions for each of the exercises.
  Interventions: Other: Clinical Based Isometric contraction strengthening Exercises using Thera band; Other: Telemonitored Home based Isometric Cntraction strengthening exercises using Thera band
- Telemonitored Home based Isometric Contraction strengthening exercises using Thera band" THB (Experimental): Participants underwent strengthening exercises to the quadriceps and harmstrings with thera band but doing the intervention at home but monitored with telephone call. The band was attached around the ankle for strengthening of the quadriceps and hamstring muscles using isometric muscle contraction using a standard protocol. The patient performed four sets of eight repetitions for each of the exercises.
  Interventions: Other: Clinical Based Isometric contraction strengthening Exercises using Thera band; Other: Telemonitored Home based Isometric Cntraction strengthening exercises using Thera band

INTERVENTIONS:
Other: Clinical Based Isometric contraction strengthening Exercises using Thera band — Patients did isometric contraction exercises using thera band in the clinic physically. They did not need to be monitored by telephone
  Other Names: Clinical Based intervention
Other: Telemonitored Home based Isometric Cntraction strengthening exercises using Thera band — Patients did isometric contraction exercises using thera band at home, they were monitored by telephone three times in a week for 8 weeks
  Other Names: Telemonitores Home based Intervention

SUMMARY:
This study assessed and compared the effects of clinic-based and telemonitored home-based interventions on pain intensity, function and quality of life in patients with knee osteoarthritis (KOA). This was with a view to providing evidence for the validation of the effectiveness of home-based intervention on knee osteoarthritis

DETAILED DESCRIPTION:
This study was a quasi-experiment involving forty two patients with KOA. They were randomly allocated into two groups equally; clinic-based group (CBG) and telemonitored home-based group (THG).

The CBG received exercises to strengthen the quadriceps and hamstring muscles using thera band while THG received same treatment regimen but at home and were monitored on phone by the researcher. The subjects performed four sets of eight repetitions for each of the exercises three days in a week for eight weeks. Pain intensity was assessed with Quadruple Visual Analog Scale, function was assessed with the Western Ontario and McMaster University Osteoarthritis Index and quality of life was assessed with WHO Quality of Life-BREF at pretreatment, 3rd week, 6th week and 8th week of intervention. Data was analysed with descriptive and inferential statistics. Repeated measure ANOVA was used to compare the mean value of variables within the group and between the groups. Alpha level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with osteoarthritis of the knee of not less than six weeks.
* Patients that have means of communication via mobile telephone.
* Patients who understands English or Yoruba Language.

Exclusion Criteria:

Participants that have any other knee joint diseases.

* Participants with history of knee joint trauma.
* Participants with history of knee surgery or arthroplasty

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
Quadruple Visual Analog Scale (QVAS) | 1-8 weeks
  This was used to assess pain intensity experienced by the participants at the time of assessment, typical or average pain, pain at its best, and pain at its worst, respectively (Von Korff et al, 1993).It consists of 4 items with each item numbered 0 to 10. With 0 indicating no pain and 10 is worst possible pain. A Yoruba translated version of the QVAS was used for participants who had preference for the Yoruba language

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index | 1-8 weeks
  WOMAC is a self-administered health-status instrument for patients with KOA, consists of 24 items within three subscales: pain (5 items), stiffness (2 items) and physical function (17 items). The Yoruba version of WOMAC translated was used for participants who do not understand English. Minimum is 0 and maxmum is 4

CONTACTS AND LOCATIONS:
Locations (1):
- Obafemi Awolowo University,, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share the IPD later

REFERENCES:
- [Background] Russell TG, Buttrum P, Wootton R, Jull GA. Internet-based outpatient telerehabilitation for patients following total knee arthroplasty: a randomized controlled trial. J Bone Joint Surg Am. 2011 Jan 19;93(2):113-20. doi: 10.2106/JBJS.I.01375. PMID 21248209
- [Background] Runhaar J, Koes BW, Clockaerts S, Bierma-Zeinstra SM. A systematic review on changed biomechanics of lower extremities in obese individuals: a possible role in development of osteoarthritis. Obes Rev. 2011 Dec;12(12):1071-82. doi: 10.1111/j.1467-789X.2011.00916.x. Epub 2011 Aug 3. PMID 21812903
- [Background] Ojoawo AO, Malomo EO, Olusegun EO, Olaogun BMO. Effects of pulse ultrasound and kneading massage in managing individual with incessant pain at lower region of back using random allocation. J Exerc Rehabil. 2018 Jun 30;14(3):516-522. doi: 10.12965/jer.1836126.063. eCollection 2018 Jun. PMID 30018942